CLINICAL TRIAL: NCT05145257
Title: Study to Evaluate the Efficacy of Elix's Cycle Balance and Its Impact on PMS and Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zenchi, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20239Elix
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: PMS; Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Masking Description: Open-label observational single-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elix Cycle Balance (Other): Elix Cycle Balance supplement
  Interventions: Dietary Supplement: Elix Cycle Balance

INTERVENTIONS:
Dietary Supplement: Elix Cycle Balance — Each day in the morning and at night in the week prior to the menstruation, the participants will take 6 full droppers of Elix Cycle Balance

SUMMARY:
This is an open-label observational single-group clinical trial to study the efficacy of a commercially available dietary supplement and its effect on common PMS and menstrual symptoms.

It is hypothesized that the dietary supplement marketed as "Elix Cycle Balance" will improve subjective wellbeing in trial participants by alleviating common symptoms of PMS and menstrual symptoms, such as cramps, bloating, and mood swings.

A total of 65 participants will be recruited for the trial following screening, with the expectation that at least 50 participants will complete the trial. The trial will be fully remote, a technology platform will be utilized to screen, enroll and capture study data of the participants. The total intervention study period will be 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-36
* Self-reported moderate to severe discomfort during menstruation, related to pelvic cramps, bloating, mood swings, or fatigue
* May experience regular or irregular menstrual cycle
* May be on birth control
* Must know or can estimate the date of the next cycle/period
* May find blood clots in menstrual blood
* Must be in good health (doesn't report any medical conditions asked in the screening questionnaire)
* Following a stable, consistent diet regimen
* Follow a stable, consistent exercise regimen and are willing, for the duration of the study, to not decrease or increase the amount of exercise in their regimen
* Agree to refrain from any lifestyle changes that may affect their menstrual cycle for the duration of the study (for example, getting on or off hormonal birth control, reducing the amount of exercise)
* Follow a stable consistent regimen when using any other interventions, such as massage, chiropractic medicine, or acupuncture; agree not to increase or decrease the number of their other interventions
* Willingness to adhere to the dietary supplement regimen
* Willingness to refrain from any other dietary supplements targeting the menstrual cycle during the study period
* Is able to communicate in English
* Is willing and able to share feedback via the used technology portal
* Must provide written informed consent (ICF)

Exclusion Criteria:

* Don't experience a menstrual cycle
* Can't estimate the onset of their next menstrual cycle
* Don't experience menstrual cramping
* Follow an extreme diet intervention
* Experienced severe weight loss in the past 3 months prior to study participation
* Usage of any medication or herbal remedies/supplements which can affect the menstrual cycle
* If currently taking allowed supplements, the dosage needs to remain the same throughout the entirety of the study
* Food intolerances/allergies that require an EpiPen
* Known allergic reaction to any of the test product ingredients
* Currently pregnant, want to become pregnant for the duration of the study, or who are breastfeeding
* Previous users of Elix Cycle Balance
* Having more than 3 alcoholic drinks a day
* Have been diagnosed with the following conditions: PCOS, Endometriosis, PMDD, Adenomyosis, Hashimoto's, anorexia, bulimia, orthorexia, binge eating, any other eating disorder
* Smokers
* Not been on a stable dose of birth control for the past 6 months

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, MSc, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Main recruitment took place between 1/5/2022 - 1/10/2022 when 65 participants were recruited. A further 3 participants were recruited on 01/26/2022.
Period: Overall Study
Arm/Group | Elix Cycle Balance
Started | 68
Completed | 61
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Survey-based assessment (0-5 scale) of menstrual symptoms [Mean (Standard Deviation); unit: units on a scale] | 4.07 (0.49)
Use of over-the-counter NSAIDS in the Treatment of Primary Dysmenorrhea Symptoms. [Mean (Standard Deviation); unit: Number of painkillers taken per day] — Survey-based assessment to assess the change in the number of over-the-counter NSAIDS used from baseline to 12 weeks. Participants were presented with the following options: 1 a day, 2 a day, 3 a day, 4+ a day. A lower score indicates a better outcome.
  Number of painkillers taken per day | 2.17 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Relief From Premenstrual Cramps [Time Frame: Baseline to 3 Months]
Description: Survey-based assessment (0-5 scale) of changes in premenstrual cramps. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.41 (1.10)
  Month 1 | 3.48 (1.18)
  Month 2 | 3.12 (1.14)
  Month 3 | 2.72 (1.09)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

2. Primary Outcome: Relief From Menstrual Cramps During the Period [Time Frame: Baseline to 3 Months]
Description: Survey-based assessment (0-5 scale) of changes in menstrual cramps. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 5.00 (0.92)
  Month 1 | 3.95 (1.31)
  Month 2 | 3.30 (1.24)
  Month 3 | 3.02 (1.30)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

3. Primary Outcome: Reduction in Usage of OTC NSAIDS in the Treatment of Primary Dysmenorrhea Symptoms. [Time Frame: Baseline to 3 Months]
Description: Survey-based assessment to assess the change in the number of over-the-counter NSAIDS used from baseline to 12 weeks. Participants were presented with the following options: 1 a day, 2 a day, 3 a day, 4+ a day. A lower score indicates a better outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: NSAID tablets per day
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
NSAID tablets per day
  Baseline | 2.05 (0.16)
  Month 1 | 1.32 (0.06)
  Month 2 | 1.07 (0.13)
  Month 3 | 0.86 (0.03)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

4. Secondary Outcome: Reduction in Mood Swings. [Time Frame: Baseline to Week 12]
Description: Survey-based assessment (0-5 scale) of changes in mood swings. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.59 (1.01)
  Month 1 | 3.36 (1.19)
  Month 2 | 3.15 (1.29)
  Month 3 | 2.75 (1.41)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

5. Secondary Outcome: Feelings of Anxiety and Depression. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in anxiety and depression. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.36 (1.20)
  Month 1 | 3.59 (1.38)
  Month 2 | 3.15 (1.40)
  Month 3 | 2.84 (1.37)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

6. Secondary Outcome: Relief From Acne Flare-ups. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in acne flare ups. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.74 (1.41)
  Month 1 | 3.02 (1.35)
  Month 2 | 2.51 (1.35)
  Month 3 | 2.33 (1.31)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

7. Secondary Outcome: Relief From Headaches. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in headaches. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.08 (1.32)
  Month 1 | 2.92 (1.40)
  Month 2 | 2.64 (1.39)
  Month 3 | 2.49 (1.27)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

8. Secondary Outcome: Relief From Backaches. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in backaches. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.15 (1.33)
  Month 1 | 3.05 (1.38)
  Month 2 | 2.62 (1.28)
  Month 3 | 2.38 (1.48)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

9. Secondary Outcome: Relief From Body Aches. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in body aches. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.67 (1.38)
  Month 1 | 2.44 (1.31)
  Month 2 | 2.28 (1.27)
  Month 3 | 2.08 (1.18)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

10. Secondary Outcome: Relief From Bloating. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in bloating. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.21 (1.22)
  Month 1 | 3.21 (1.21)
  Month 2 | 2.87 (1.29)
  Month 3 | 2.51 (1.36)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

11. Secondary Outcome: Relief From Gastrointestinal Issues. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in gastrointestinal issues. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.97 (1.38)
  Month 1 | 3.05 (1.51)
  Month 2 | 2.74 (1.25)
  Month 3 | 2.26 (1.29)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

12. Secondary Outcome: Relief From Joint or Muscle Pain. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in joint or muscle pain. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.46 (1.52)
  Month 1 | 2.31 (1.30)
  Month 2 | 2.16 (1.05)
  Month 3 | 1.90 (1.10)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

13. Secondary Outcome: Relief From Tiredness or Fatigue. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in tiredness and fatigue. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 4.69 (0.96)
  Month 1 | 3.62 (1.20)
  Month 2 | 3.26 (1.39)
  Month 3 | 2.93 (1.30)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

14. Secondary Outcome: Reduction in Weight Gain Due to Fluid Retention. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in menstrual symptoms, fatigue, and mood swings. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.49 (1.51)
  Month 1 | 2.66 (1.40)
  Month 2 | 2.31 (1.27)
  Month 3 | 2.08 (1.27)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

15. Secondary Outcome: Relief From Breast Tenderness. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in breast tenderness. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.30 (1.41)
  Month 1 | 2.62 (1.38)
  Month 2 | 2.20 (1.30)
  Month 3 | 1.93 (1.18)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

16. Secondary Outcome: Changes in Appetite and Food Cravings. [Time Frame: Baseline to Month 3]
Description: Survey-based assessment (0-5 scale) of changes in appetite and food cravings. On the scale, 0 = "No symptoms" and 5 = "Severe It interferes with my daily life, and I cancel activities". Lower scores indicate a favourable outcome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elix Cycle Balance
Number analyzed (Participants) | 61
score on a scale
  Baseline | 3.98 (1.20)
  Month 1 | 3.03 (1.31)
  Month 2 | 2.31 (1.21)
  Month 3 | 2.16 (1.13)
Statistical Analysis 1: Comparison: Elix Cycle Balance; Test type: Other; p < 0.001, ANOVA — Baseline versus endline comparison

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial. Each participant was monitored for the 3 months they took part in the trial.
Description: All participants were monitored for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Elix Cycle Balance
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 7/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elix Cycle Balance (N=68)
Stomach upset (Gastrointestinal disorders) | 1 (1) — One participant withdrew from the trial due to stomach upset.
Headache (General disorders) | 1 (1) — One participant withdraw from the trial due to headaches.
Personal Issue (Social circumstances) | 1 (1) — One participant withdrew from the trial due to a personal issue unrelated to the product.
No response (Product Issues) | 4 (4) — Four participants withdrew from the trial as they reported nil effect or response from the product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT05145257/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT05145257/ICF_001.pdf